CLINICAL TRIAL: NCT06918574
Title: The Effect of Breastfeeding Roadmap on Breastfeeding Self-Efficacy Perception and Breastfeeding Success in Primiparous Women
Brief Title: Breastfeeding Roadmap in Primiparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ebru Bekmezci, PhD, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/048
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breastfeeding; Self Efficacy
Keywords: Breastfeeding Roadmap
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to the routine breastfeeding education given by the clinic's education nurse, the mothers in the intervention group will also receive a "Breastfeeding Roadmap" education poster prepared by the researchers, which will be hung on the wall of their rooms. The researcher will introduce the Breastfeeding Roadmap to the mothers and provide information on breastfeeding.
  Interventions: Other: Breastfeeding Education with Breastfeeding Roadmap
- Control group (No Intervention): The control group of the study will receive routine breastfeeding education provided by the clinic's education nurse.

INTERVENTIONS:
Other: Breastfeeding Education with Breastfeeding Roadmap — Information about the "Breastfeeding Roadmap" prepared by the researchers will be explained to the mothers in the intervention group and hung in poster rooms.
  Arms: Intervention group

SUMMARY:
The effect of the breastfeeding roadmap used in primiparous mothers on breastfeeding self-efficacy perception and breastfeeding success will be evaluated.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled experimental study. Mothers who meet the inclusion criteria and agree to participate in the study will be assigned to the intervention and control groups according to the randomization list.

A total of 74 primiparous mothers who gave birth, 37 in the intervention group and 37 in the control group, will be included in the study.

In addition to the routine breastfeeding education given by the clinic's education nurse, the mothers in the intervention group will also receive a "Breastfeeding Roadmap" education poster prepared by the researchers, which will be hung on the wall of their rooms. The researcher will introduce the Breastfeeding Roadmap to the mothers and provide information on breastfeeding. Routine hospital breastfeeding education will receive to mothers in the control group after childbirth.

Data Collection Pre-Test; Introductory Information Form, Breastfeeding Self-Efficacy Scale Short-Form, LATCH Breastfeeding Assessment Tool will be collected within the first hour after birth (before Breastfeeding Roadmap breastfeeding education and hospital routine breastfeeding education were implemented) Post-test; Breastfeeding Self-Efficacy Scale Short-Form, LATCH Breastfeeding Assessment Tool will be collected at least two hours before mothers are discharged from the hospital (the discharge period usually varies between 24 and 48 hours).

At the end of the study, the results of the mothers in the experimental and control groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* Primiparous,
* Giving birth at 37 weeks of gestation or later,
* No condition preventing breastfeeding,
* No condition preventing breastfeeding in the baby,
* At least primary school graduate,
* Mothers aged 18 and over

Exclusion Criteria:

* Those who have given birth to multiple pregnancies,
* Those who received general anesthesia for Caesarean section,
* Those who have any chronic disease, diagnosed mental or psychiatric illness history,
* Those who have a history of preeclampsia, eclampsia and gestational diabetes,
* Those whose babies are in intensive care after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Sociodemographic characteristics | Within the first hour after the mother's birth.
  Comparison of sociodemographic characteristics of women before the intervention with the questionnaire
Breastfeeding Self-Efficacy Short Form Scale | Within the first hour after the mother's birth.
  Mothers whose pre-test data are collected will be assigned to intervention and control groups (Pre-test).
  The scale consists of 14 items. It is scored between 1-5 and the lowest 14 and the highest 70 points can be obtained. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Self-Efficacy Short Form Scale | At least two hours before mothers are discharged from the hospital (the discharge period usually varies between 24 and 48 hours)
  Post-test data will be collected before mothers are discharged from the hospital (Post-test).
  The scale consists of 14 items. It is scored between 1-5 and the lowest 14 and the highest 70 points can be obtained. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
LATCH Breastfeeding Assessment Tool | Within the first hour after the mother's birth
  Mothers whose pre-test data are collected will be assigned to intervention and control groups (pre-test).
  The scale consists of five evaluation criteria and each item is evaluated between 0-2 points. The score that can be obtained from the measurement tool can vary between 0-10. The higher the score obtained from the scale, the higher the breastfeeding success.
LATCH Breastfeeding Assessment Tool | At least two hours before mothers are discharged from the hospital (the discharge period usually varies between 24 and 48 hours)
  Post-test data will be collected before mothers are discharged from the hospital (Post-test).
  The scale consists of five evaluation criteria and each item is evaluated between 0-2 points. The score that can be obtained from the measurement tool can vary between 0-10. The higher the score obtained from the scale, the higher the breastfeeding success.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Bekmezci PhD, Principal Investigator — Selcuk University; Hediye Karakoç PhD, Principal Investigator — KTO Karatay University; Halime Esra Meram PhD, Principal Investigator — Selcuk University; Jule Eriç Horasanlı Doctor, ASSOCIATE PROFESSOR, Principal Investigator — Necmettin Erbakan University Medical Faculty Hospital
Locations (1):
- Necmettin Erbakan University Faculty of Medicine Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No